CLINICAL TRIAL: NCT02592629
Title: The Efficacy of Local Anesthetics to Reduce Shoulder Pain Post-Steroid Injections
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of time to enroll due to additional responsibilities of the PI and research coordinator.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Robert A. Gallo, Assistant Professor of Surgery Orthopaedics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2690
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Shoulder Pain
Keywords: subacromial injection; rotator cuff disease; steroid injection
MeSH Terms: conditions — Shoulder Pain | interventions — Lidocaine; Ethyl Chloride; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- no topical or subcutaneous anesthetic (Active Comparator): Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine
  Interventions: Drug: lidocaine; Drug: Kenalog
- subcutaneous lidocaine (Active Comparator): Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine after 2 ml or 1% lidocaine by subcutaneous injection
  Interventions: Drug: lidocaine; Drug: Kenalog
- topical ethyl chloride (Active Comparator): Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine after applying ethyl chloride spray for 3 seconds
  Interventions: Drug: lidocaine; Drug: ethyl chloride; Drug: Kenalog

INTERVENTIONS:
Drug: lidocaine — used with Kenalog in shoulder injection and as topical anesthetic as subcutaneous injection
  Other Names: xylocaine
Drug: ethyl chloride — topical spray
  Other Names: chloroethane
  Arms: topical ethyl chloride
Drug: Kenalog — used with lidocaine in shoulder injection
  Other Names: triamcinolone

SUMMARY:
The specific aim of this prospective study is to determine whether local anesthetics prior to subacromial steroid injections reduce pain and consequently if they are cost-effective in the treatment for shoulder pathology.

DETAILED DESCRIPTION:
Shoulder pain is a common problem that can be estimated to be prevalent in up to 15 percent of the patient population registered to general practices and is second only to back pain in patients seeking treatment for musculoskeletal issues in the primary care setting. As a common source of distress, shoulder pain contributes significantly to health care costs.

Rotator cuff disease due to impingement, tendonitis or bursitis is a frequent cause of shoulder pain and dysfunction. Initial treatment consists of a conservative approach of activity modification, oral nonsteroidal anti-inflammatory drugs (NSAIDs) and supervised physical therapy. However, if the patients' symptoms persist, subacromial injections of a local anesthetic such as lidocaine, and a corticosteroid may be indicated as a sequential treatment option.

The steroid injection itself can be a painful process, so administering a local anesthetic prior to the steroid injection is thought to mitigate pain or reduce possible discomfort during and immediately following the procedure. Though there is evidence advocating for the benefits of combining local anesthetics and corticosteroids for the treatment of subacromial pathologies, it is not conclusive whether local anesthesia significantly enhances the pain relieving effect of steroids. Should local anesthesia not have a significant impact on the patient's pain intensity, then the use of corticosteroids alone could potentially result in reduced costs in care.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 70 years old
* Shoulder pain lasting at least 4 weeks
* Inability to use arm with restriction of movement and loss of full function.
* Able to understand study and provide voluntary, written informed consent

Exclusion Criteria:

* Less than 18 or greater than 70 years old
* Contraindications of previous injections and previous shoulder surgery
* Unable to understand consent form (in the opinion of the PI)
* Non-English speaking individuals
* Medication contradictions to lidocaine, corticosteroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Gallo, MD, Principal Investigator — The Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | no Topical or Subcutaneous Anesthetic | Subcutaneous Lidocaine | Topical Ethyl Chloride
Started | 5 | 9 | 5
Completed | 5 | 9 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | no Topical or Subcutaneous Anesthetic | Subcutaneous Lidocaine | Topical Ethyl Chloride | Total
Number analyzed (Participants) | 5 | 9 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 5 | 19
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 2 | 12
  Male | 2 | 2 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 9 | 5 | 19
baseline pain [Mean (Standard Deviation); unit: units on a scale] — The pain will be measured with a scale from 0 (no pain) to 10 (worst possible pain)".
  units on a scale | 4.2 (2.56) | 5.16 (1.93) | 4.7 (1.84) | 4.78 (2.11)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Assessment
Description: Pain assessed on a visual analog scale from 1 (no pain) to 10 (worst pain imaginable). Pain score at 10 minutes post-injection is subtracted from baseline pre-injection score. Positive numbers to represent increases and negative numbers to represent decreases.
Time Frame: change from baseline assessment before injection at 10 minutes post injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Topical or Subcutaneous Anesthetic | Subcutaneous Lidocaine | Topical Ethyl Chloride
Number analyzed (Participants) | 5 | 9 | 5
units on a scale | 3 (1.6) | 4.21 (2.19) | 5.6 (1.88)
Statistical Analysis 1: Comparison: no Topical or Subcutaneous Anesthetic vs Subcutaneous Lidocaine vs Topical Ethyl Chloride; Test type: Equivalence — ANOVA; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | no Topical or Subcutaneous Anesthetic | Subcutaneous Lidocaine | Topical Ethyl Chloride
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT02592629/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT02592629/Prot_SAP_001.pdf